CLINICAL TRIAL: NCT04182971
Title: Effect of Added Fruit Pomace Fiber, Juice, and Whole Fruit on Postprandial Glycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1806
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Glycemic Index
Keywords: Juice; Fiber
MeSH Terms: interventions — Fruit; Fruit and Vegetable Juices; Dietary Fiber

STUDY DESIGN:
Intervention Model Description: Cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole fruit (Active Comparator): Phase 1 of study is an orange, Phase 2 of study is an apple
  Interventions: Other: Fruit
- Juice (Active Comparator): Phase 1 of study is orange juice, Phase 2 of study is apple juice
  Interventions: Other: Fruit juice
- Juice plus pomace fiber (Experimental): Phase 1 is orange juice with added fiber, Phase 2 is apple juice with added fiber
  Interventions: Other: Fruit juice plus fiber

INTERVENTIONS:
Other: Fruit — Phase 1 is 227g of orange fruit, Phase 2 is 230g of apple fruit
  Arms: Whole fruit
Other: Fruit juice — Phase 1 is 250g of orange juice, Phase 2 is 235g of apple juice
  Arms: Juice
Other: Fruit juice plus fiber — Phase 1 is 157g of orange juice + 100g of orange pomace fiber (39% pomace by weight), Phase 2 is 129g of apple juice + 106g of apple pomace fiber (45% pomace by weight)
  Arms: Juice plus pomace fiber

SUMMARY:
Compare the effects of whole orange, orange juice alone, and orange juice with added orange pomace fiber, and whole apple, apple juice alone, and apple juice with added apple pomace fiber, on 2h glycemic response.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-24.9 kg/m2 and weight >=110 lbs at screening
* Willing to maintain usual physical activity pattern and exercise level
* Willing to follow instructions for compliance with dietary restrictions, dosing and visits
* In good health based on medical history
* Willing to avoid alcohol for 24 hrs prior to visits
* Willing to maintain stable dose of vitamins, minerals, supplements, and medications not interfering with study outcomes including birth control for the study
* Understands procedures, signs informed consent and authorization for release of relevant protected health information and is willing to complete study procedures

Exclusion Criteria:

* Fasting finger stick glucose >100
* Uncontrolled hypertension
* Major trauma or surgical event within 2 months of Visit 1
* Weight change > 4.5 kg within 2 months, taking weight loss drugs, bariatric surgery, or other weight reduction surgery (liposuction, laser fat removal, etc.)
* History or presence of clinically important endocrine, cardiovascular, pulmonary, bilary or gastrointestinal disorders that could interfere with the interpretation of study results
* History or presence of cancer in past 2 yrs except for non-melanoma skin cancer
* History of extreme dietary habits (Atkins, etc.)
* History of eating disorder
* Known intolerance or sensitivity to any of the ingredients in the study products
* Subject has used medications know to influence carbohydrate metaboism 2 weeks prior to visit and throughout the study
* Subject is taking systemic steroids, extreme alcohol use or drug user
* Vein access score < 7
* Pregnant, planning to become pregnant, or lactating
* Current smoker or smoked within past 2 yrs
* Has not participated in another clinical trial for past 30 days or another PepsiCo study in past 6 months

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Glucose | 0-120 minutes
  Cmax, plasma

SECONDARY OUTCOMES:
Glucose | 0-120 minutes
  iAUC, plasma
Insulin | 0-120 minutes
  iAUC, plasma
Glucose | 0-120 minutes
  Tmax, plasma
Insulin | 0-120 minutes
  Cmax, plasma
Insulin | 0-120 minutes
  Tmax, plasma

CONTACTS AND LOCATIONS:
Locations (1):
- IIT (Illinois Institute of Technology), Center for Nutrition Research, Institute for Food Safety and Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
After publication, investigator can be contacted to discuss requests.